CLINICAL TRIAL: NCT06519526
Title: Exploratory Clinical Study of SHR-0302 and SHR-2554 in Patients With Relapsed/Refractory Peripheral T Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Rong Tao, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTCL-IIT-SHR2554-SHR0302
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Relapsed/Refractory Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — ivarmacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-0302 and SHR-2554 Treatment Arm (Experimental): SHR-2554 Oral administration, twice daily, with a 28-day continuous dosing as one cycle. SHR-0302: Oral administration, once daily,
  Interventions: Drug: SHR-0302; Drug: SHR-2554

INTERVENTIONS:
Drug: SHR-0302 — SHR-0302 will be administered orally as tablets.
Drug: SHR-2554 — SHR-2554 will be administered orally as tablets.

SUMMARY:
This is an open-label, prospective and exploratory clinical study to evaluate the efficacy and safety of JAK inhibitor SHR-0302 in combination with EZH2 inhibitor SHR-2554 in patients with R/R PTCL. The study plans to enroll approximately 25 patients. 6-12 patients will receive SHR-0302 monotherapy and SHR-0302+SHR-2554 combination therapy in the safety run-in phase. According to the safety observed, the investigators discuss and decide to select a dose group to explore the efficacy and safety. 13 patients may be enrolled in the expansion phase.

DETAILED DESCRIPTION:
This is an open-label, prospective, exploratory clinical study. The plan is to enroll 12-25 patients with relapsed/refractory peripheral T-cell lymphoma (r/r PTCL) to receive a combination of SHR-0302 and SHR-2554. The primary objectives are to evaluate the efficacy and safety of the SHR-0302 and SHR-2554 combination in the treatment of r/r PTCL. Subjects will receive the investigating drugs combination (SHR-0302 and SHR-2554) until study completion, unacceptable toxicity, disease progression, withdrawal of informed consent, or investigators discontinue treatment.

The study is divided into two parts. Part I is a safety run-in phase, and part II is an efficacy exploration phase.

Part I:

Cohort 1: Explore the recommended dose and safety of SHR-0302 monotherapy Cohort 2: Based on the efficacy and safety observed in Cohort 1, explore the clinically recommended dose and safety of the SHR-0302 and SHR-2554.

Part II: Based on the safety and tolerability observed during part I, the investigators will discuss and select one tolerable dose cohort to explore the efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18-70 years (inclusive);
* Histologically confirmed peripheral T-cell lymphoma;
* Disease status defined as relapsed or refractory after >=1 prior systemic treatment lines;
* Have measurable lesions;
* ECOG performance status must be 0 or 1 and has not deteriorated in the past 2 weeks;
* Life expectancy ≥12 weeks;
* Adequate bone marrow reserve and organ system function reserve;
* Participants should be able and willing to comply with the study protocol requirement;

Exclusion Criteria:

* Received anti-tumor treatment within 28 days prior to the first dose of the study drug; received Chinese medicine treatment with anti-tumor effect within 14 days before the first dose of the study drug; received steroid hormones within 7 days prior to the first dose of study drug administration;
* Underwent major surgery within 4 weeks prior to the first dose of study treatment；
* Severe cardiovascular disease;
* Cerebrovascular accident or transient ischemic attack within 6 months prior to enrollment;
* Significant impairment of lung function;
* Active infections;
* Unexplained fever > 38.5°C during screening period or on the first day of medication;
* Pregnant;
* Known alcohol or drug abuse;
* Subjects are currently receiving known moderately potent or potent CYP inducers/inhibitors or P-glycoprotein (P-gp) inhibitors;
* History of hypersensitivity to the investigational drug or its excipients;
* In the judgment of the investigator, objective conditions make the subject unable to complete the planned study or the subject has other factors, concomitant diseases, combined treatment or abnormal laboratory examination that may lead to the forced termination of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of AEs and SAEs | The first dose until 30 days after last dose
  Incidence and severity of AEs and SAEs will be recorded and graded according to the CTCAE 5.0.
Objective response rate (ORR) | 24 months
  Percentage of participants achieving complete response (CR) and partial response (PR) according to Lugano 2014 criteria.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 24 months
  Percentage of patients achieving complete response (CR) and partial response (PR) and stable disease (SD) according to Lugano 2014 criteria.
Duration of Response (DoR) | 24 months
  Defined as the time from the date of the first CR or PR to the date of the first PD or death due to any cause, whichever occurs first.
Progression-free Survival (PFS) | 24 months
  Defined as the time from the date of the first dose to the first documented PD or death due to any cause, whichever occurs first.
Overall Survival (OS) | 24 months
  Defined as the duration of time from start of treatment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Rong Tao, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China